CLINICAL TRIAL: NCT00600600
Title: Use of Tigecycline for Treatment of Serious Infection Due to Rapidly Growing Mycobacteria (Especially M.Abscessus)
Brief Title: Tigecycline for Treatment of Rapidly Growing Mycobacteria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at Tyler (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Richard J. Wallace, Jr., M.D., Chairman Department of Microbiology, The University of Texas Health Science Center at Tyler
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 660
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Mycobacterium Abscessus Lung Disease; Rapidly Growing Mycobacterial Lung Disease
MeSH Terms: interventions — Tigecycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tigecycline (Experimental): tigecycline titrated dose according to patient age and clinical status
  Interventions: Drug: Tigecycline

INTERVENTIONS:
Drug: Tigecycline — Tigecycline dosage based on age and clinical status of patient.
  Other Names: tygacil

SUMMARY:
To determine the safety, tolerance, and efficacy of Tigecycline when given daily to patients with rapidly growing mycobacterial disease (especially M.abscessus).

DETAILED DESCRIPTION:
To assess the safety and efficacy of tigecycline in the treatment of drug resistant rapidly growing mycobacterial disease especially M. abscessus

ELIGIBILITY:
Inclusion Criteria:

* Positive cultures for rapidly growing mycobacteria
* Patients who have drug resistant isolates or are intolerant of macrolides or have serious infections unresponsive to currently available drugs
* Adults and children 10 years of age and older
* Pretreatment isolate of M. avium complex available for MIC determination
* Available for followup appointments

Exclusion Criteria:

* History of tetracycline allergy
* If a menstruating female, not pregnant and on adequate birth control

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2002-04; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical and microbiological outcomes such as clinical symptoms and laboratory cultures | 6 mos
  culture neg X3 ( sputum conversion)

SECONDARY OUTCOMES:
clinical and Microbiological outcomes | 6 mos
  clinical and radiographic improvements

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Wallace Jr., M.D., Principal Investigator — The University of Texas Health Science Center at Tyler
Locations (1):
- The University of Texas Health Science Center at Tyler, Tyler, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallace RJ Jr, Dukart G, Brown-Elliott BA, Griffith DE, Scerpella EG, Marshall B. Clinical experience in 52 patients with tigecycline-containing regimens for salvage treatment of Mycobacterium abscessus and Mycobacterium chelonae infections. J Antimicrob Chemother. 2014 Jul;69(7):1945-53. doi: 10.1093/jac/dku062. Epub 2014 Mar 14. PMID 24633206